CLINICAL TRIAL: NCT01536353
Title: A Single Dose, Randomized, Open-label, 2x2 Crossover Study to Evaluate the Bioavailability and Safety of AGSAV301 Tablet in Healthy Male Volunteers
Brief Title: Clinical Trial to Evaluate the Bioavailability and Safety of AGSAV301
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1110-AGSAV-P1
Record Dates: First submitted 2012-02-15; First posted 2012-02-22 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (2):
- AGSAV301 (Experimental)
  Interventions: Drug: AGSAV301
- Exforge 10/160 (Active Comparator)
  Interventions: Drug: Exforge 10/160

INTERVENTIONS:
Drug: AGSAV301 — tablet, q.d.
  Arms: AGSAV301
Drug: Exforge 10/160 — Tablet, q.d.
  Arms: Exforge 10/160

SUMMARY:
The purpose of this study is to evaluate the bioavailability and safety of AGSAV301 tablet in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 20 to 40 years at screening.
* body weight ≥ 45kg and within ± 20% of the ideal body weight : Ideal body weight = (height [cm] - 100) x 0.9
* Be able to collect blood for study and visit for follow-up period
* Subject who agrees to participate in this study and give written informed consent

Exclusion Criteria:

* Have history of significant hepatic, renal, gastrointestinal, pulmonary, musculoskeletal, endocrine, neuropsychiatric, hematologic, cardiovascular diseases
* Have a gastrointestinal disease(ex : Crohn's disease, gastrointestinal ulcer)or surgery(except for Appendectomy, Hernia repair) affected the absorption of medications
* Inappropriate in Screening test (interview, vital sigh, BP, 12-lead ECG, laboratory test etc.)
* Hypersensitivity reactions to drugs or clinically significant hypersensitivity reactions in the history of amlodipine or valsartan
* drug abuse, or have a history of drug abuse showed a positive for the screening test on urine : amphetamine, barbiturate, cocaine, opiates, benzodiazepines, cannabinoids, methadone etc.
* Subject who takes herbal medicine within 30 days, ethical drug within 14 days, OTC within 7 days before the beginning of administration of investigational drug
* Unusual diet affected the absorption, distribution, metabolism, excretion of medications
* Subject who treated with any investigational drugs within 60 days before the administration of investigational drug
* Previously donate whole blood within 60 days or component blood within 30 days or transfusion within 30 days
* Subject who takes inhibitors and inducers of drug metabolizing enzyme (Barbiturates etc.) within 30days
* Subject who have taken habitually caffeine (caffeine > 5 units/day)
* Subject who have drunken habitually (alcohol > 21 units/week, 1 unit = pure alcohol 10ml)or who are unable to quit drinking during this study or smoker
* positive for Hepatitis B, Hepatitis C, HIV or Syphilis
* Blood Pressure is not in the range of "140 > sitting SBP ≥ 90mmHg, 90 > sitting DBP ≥ 60mmHg"
* Pulse rate is not in the range of "95 > sitting Pulse Rate ≥ 45bpm (beats per minute)"
* AST, ALT, total bilirubin over twice of reference range
* Subjects deemed ineligible by investigator based on other reasons

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 ,12, 16, 24, 36, 48, 72, 96, 120, 168 hours
Cmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 ,12, 16, 24, 36, 48, 72, 96, 120,168 hours

SECONDARY OUTCOMES:
AUC (inf) | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 ,12, 16, 24, 36, 48, 72, 96, 120,168 hours
tmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 ,12, 16, 24, 36, 48, 72, 96, 120, 168 hours
t(1/2β) | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 ,12, 16, 24, 36, 48, 72, 96, 120, 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea